CLINICAL TRIAL: NCT00748397
Title: An Open, Prospective, Multicenter Study to Evaluate Treatment of Edentulous Upper Jaws With Fixed Detachable Bridges Retained by Astra Tech Dental Implants, Fixture Micro-Macro
Brief Title: Evaluation of Treatment With Fixture Microthread™ in Patients Missing All Teeth in the Upper Jaw, When Using One-Stage Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision to modify the product under study as a result of feedback regarding subjective feeling during installation procedure. For more info, see brief summary.
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Head of Therapeutic Area Dental, Clinical Research, Astra Tech AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-MMF-0002
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Jaw, Edentulous
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Fixture MicroThread (Micro-Macro)

INTERVENTIONS:
Device: Fixture MicroThread (Micro-Macro) — Fixture MicroThread (Micro-Macro) Ø 3.5 and 4.0 mm in lengths of 9, 11, 13, 15 and 17 mm.

SUMMARY:
The primary objective of the study is to evaluate the long-term survival rate of implants and prostheses when treating totally edentulous upper jaws with Fixture MicroThread (Micro-Macro) using a one-stage surgical procedure.

Clinical study recruitment was stopped in year 2000 due to a decision to modify the product under study. This was a result of feedback regarding the subjective feeling during the installation procedure. There were no safety concerns w/r to the study products. Patients already included and treated in the study were monitored for the full duration of the study in accordance with the clinical study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Sufficient amount of bone to give good support for implants of at least 9 mm length.
* Willing to give signed informed consent

Exclusion Criteria:

* Any systemic disease or condition that would compromise post-operative healing and/or osseointegration
* Systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Unable or unwilling to return for follow-up visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1999-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Implant survival | Continuously during 5,5 years after implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Bo Sunzel, Dr, Principal Investigator — Käkkirurgiska kliniken, Universitetssjukhuset MAS
Locations (4):
- Louisiana State University Medical Center, School of Dentistry, New Orleans, Louisiana, United States
- Klinik und Poliklinik fur Mund- Kiefer- und Geschichtechirurgie, Ruprecht-Karls-Universität, Heidelberg, Germany
- Dpto. Medicina y Cirugia Bucofacial, Facultad de Odontologia, Madrid, Spain
- Käkkirurgiska kliniken, Universitetssjukhuset MAS, Malmo, Sweden